CLINICAL TRIAL: NCT01326637
Title: A Human Factors Intervention to Reduce Risk in Primary Care of the Elderly
Brief Title: Human Factors Intervention to Reduce Risk in Primary Care of the Elderly
Acronym: SAFE-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010-0447; R18HS017899 (AHRQ)
Record Dates: First submitted 2011-03-23; First posted 2011-03-31 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Primary Health Care; Aged; Clinical Information
Keywords: primary health care; aged

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): Received the intervention: previsit planning phone call with filled out patient overview document & clinician huddle
  Interventions: Other: Patient Overview Document
- observation (No Intervention): Received usual care

INTERVENTIONS:
Other: Patient Overview Document — The Intervention has two components:
  1. Pre-visit care coordination:
     * 5-7 days prior to a study patient's appointment with the doctor, the doctor's nurse/MA will call the study patient and collect pertinent clinical information using a data collection form we call a Patient Overview Document or POD. The purpose of the POD is to comprehensively inform the doctor about the patient before the doctor enters the exam room.
     * The nurse/MA will ensure that lab results, consultant reports, ER reports, imaging studies, etc., needed by the physician during the patient's visit, are available to the doctor in their usual place.
  2. Team Meeting:
  On the day of the patient's appointment, prior to the beginning of the clinic session, the nurse/MA and doctor will jointly review the POD.
  Arms: intervention

SUMMARY:
Human factors engineering literature makes clear that appropriate, well-designed and well-timed information improves decision making and can reduce mental workload. Data from a previous study showed that appropriate, well-designed and well-timed information is not present in many primary care encounters with elderly patients. This puts primary care physicians at risk of higher mental workload and poor decision making which can affect the quality and safety of care delivered to patients. Elderly patients are at particular risk because they are more likely to have more comorbidities, medications, and cognitive impairments.

Dr. Karsh and his research team will test an intervention to improve the performance of primary care physicians and, thus the safety of primary care of the elderly. The investigators will use a randomized experiment, with random assignment at the level of patient, to test and evaluate the intervention. The evaluation will involve 4 primary care clinics, with 4 primary care physicians per clinic. The investigators will collect data from 768 patient visits pre-intervention and 1536 patient visits during the intervention. Intervention patients will be randomly assigned to the intervention or care as usual.

The Intervention has two components:

Pre-visit care coordination:

* 5-7 days prior to a study patient's appointment with his/her doctor, the doctor's nurse/MA will call the study patient and collect pertinent clinical information about the patient using a data collection form the investigators call a Patient Overview Document or POD.
* The nurse/MA will ensure that any lab results, consultant reports, ER reports, imaging studies, etc., that will be needed by the physician are available to the doctor.

Team Meeting:

On the day of the patient's appointment and prior to the beginning of the clinic session, the nurse/MA will meet briefly with the doctor to jointly review the POD.

Hypotheses:

H1. Primary Care Physician (PCP): The intervention will increase situation awareness, reduce PCP mental workload, reduce PCP perceived likelihood of error, and improve PCP visit satisfaction. PCP efficiency, as measured by encounter problem density during a visit, will also improve.

H2. Patient: The intervention will improve patients' perceptions of their visits on a variety of AHRQ CAHPS measures, such as physician knowledge of patient history.

H3. Patient: The intervention will not impact the number or types of problems addressed during the visit.

H4. Clinic: The intervention will not affect visit RVUs

ELIGIBILITY:
Inclusion Criteria:

* Must be greater than or equal to 65 years of age
* Must be patients of participating physicians

Exclusion Criteria:

* Cannot speak English
* Cannot hear well enough to respond to questions via the telephone or do not have a caregiver who can respond to questions on their behalf

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2332 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Number and types of problems discussed during visit | 04/12
  There are no outcome measures for individual patients.
  We will review the dictated clinic note for each study patient visit in order to
  * Make a list of the all problems (e.g., hypertension, asthma, annual influenza vaccination, etc.) that are discussed in the clinic note;
  * Record the number of problems that the patient and doctor discussed.
  We will compare the number of problems and the kind of problems found in the intervention patient group with the number and kind of problems found in the care-as-usual group.

SECONDARY OUTCOMES:
Resource utilization | 04/12
  There are no outcome measures for individual patients. We will look at the resource utilization (RVUs) during care-as-usual visits compared to resource utilization during intervention visits. To assess resource utilization, we will collect E&M/CPT codes for each study visit and calculate the RVUs. A study patient is seen only once.

CONTACTS AND LOCATIONS:
Overall Officials: Ben-Tzion Karsh, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States